CLINICAL TRIAL: NCT03985410
Title: A Randomized, Three Period Crossover Thorough QT (TQT) Study Evaluating the Effect of ETX2514 on Cardiac Repolarization in Healthy Male or Female Volunteers
Brief Title: Study Evaluating the Effect of ETX2514 on Cardiac Repolarization in Healthy Male or Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Entasis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CS2514-2018-0003
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Acinetobacter Baumannii-calcoaceticus Complex Infections
Keywords: Acinetobacter baumannii-calcoaceticus; complex infections; ETX2514; cardiac repolarization; heart rate-corrected QT interval (QTc)
MeSH Terms: interventions — durlobactam; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The administration of ETX2514 and ETX2514 placebo will be double-blinded. Placebo and moxifloxacin (Treatment Period C) will be administered open-label.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment Sequence ABC (Experimental): Participants will receive a single 3-hour intravenous (IV) infusion of 4 grams (g) of ETX2514 (supratherapeutic dose) (Treatment A), followed by a single 3-hour IV infusion of placebo for ETX2514 (Treatment B), followed by a single 3-hour IV infusion of placebo for ETX2514 and a single oral dose of 400 milligrams (mg) open-label moxifloxacin given at the end of the infusion (Treatment C). There will be 7 ± 2 days washout between treatments.
  Interventions: Drug: ETX2514; Drug: Placebo; Drug: moxifloxacin
- Treatment Sequence ACB (Experimental): Participants will receive a single 3-hour IV infusion of 4 g of ETX2514 (supratherapeutic dose) (Treatment A), followed by a single 3-hour IV infusion of placebo for ETX2514 and a single oral dose of 400 mg open-label moxifloxacin given at the end of the infusion (Treatment C), followed by a single 3-hour IV infusion of placebo for ETX2514 (Treatment B). There will be 7 ± 2 days washout between treatments.
  Interventions: Drug: ETX2514; Drug: Placebo; Drug: moxifloxacin
- Treatment Sequence BAC (Experimental): Participants will receive a single 3-hour IV infusion of placebo for ETX2514 (Treatment B), followed by a single 3-hour IV infusion of 4 g of ETX2514 (supratherapeutic dose) (Treatment A), followed by a single 3-hour IV infusion of placebo for ETX2514 and a single oral dose of 400 mg open-label moxifloxacin given at the end of the infusion (Treatment C). There will be 7 ± 2 days washout between treatments.
  Interventions: Drug: ETX2514; Drug: Placebo; Drug: moxifloxacin
- Treatment Sequence BCA (Experimental): Participants will receive a single 3-hour IV infusion of placebo for ETX2514 (Treatment B), followed by a single 3-hour IV infusion of placebo for ETX2514 and a single oral dose of 400 mg open-label moxifloxacin given at the end of the infusion (Treatment C), followed by a single 3-hour IV infusion of 4 g of ETX2514 (supratherapeutic dose) (Treatment A). There will be 7 ± 2 days washout between treatments.
  Interventions: Drug: ETX2514; Drug: Placebo; Drug: moxifloxacin
- Treatment Sequence CAB (Experimental): Participants will receive a single 3-hour IV infusion of placebo for ETX2514 and a single oral dose of 400 mg open-label moxifloxacin given at the end of the infusion (Treatment C), followed by a single 3-hour IV infusion of 4 g of ETX2514 (supratherapeutic dose) (Treatment A), followed by a single 3-hour IV infusion of placebo for ETX2514 (Treatment B). There will be 7 ± 2 days washout between treatments.
  Interventions: Drug: ETX2514; Drug: Placebo; Drug: moxifloxacin
- Treatment Sequence CBA (Experimental): Participants will receive a single 3-hour IV infusion of placebo for ETX2514 and a single oral dose of 400 mg open-label moxifloxacin given at the end of the infusion (Treatment C), followed by a single 3-hour IV infusion of placebo for ETX2514 (Treatment B), followed by a single 3-hour IV infusion of 4 g of ETX2514 (supratherapeutic dose) (Treatment A). There will be 7 ± 2 days washout between treatments.
  Interventions: Drug: ETX2514; Drug: Placebo; Drug: moxifloxacin

INTERVENTIONS:
Drug: ETX2514 — intravenous infusion
Drug: Placebo — intravenous infusion
Drug: moxifloxacin — oral tablet

SUMMARY:
This study is being conducted to evaluate the effects of supratherapeutic ETX2514 plasma concentrations on the heart rate-corrected QT interval (QTc).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, 18-55 years of age, inclusive, at Screening
* Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dose
* Must weigh at least 60 kilograms (kg) for males or 52 kg for females and have a body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/meters squared (m^2) at Screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or electrocardiograms (ECGs), as deemed by the Principal Investigator (PI)
* Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must have a negative serum pregnancy test before randomization. Participating heterosexual women of childbearing potential must be willing to consistently use 2 highly effective methods of contraception (i.e., condom with spermicide, combined oral contraceptive, implant, injectable, indwelling intrauterine device, or a vasectomized partner) from Screening until at least 30 days after administration of the last dose of study drug; and
* Non-childbearing women must have had a hysterectomy, surgical sterilization, or be postmenopausal at least 12 months prior to Screening.
* Male participants must be willing to use condoms with spermicide during sexual intercourse from Screening until at least 90 days after administration of the last dose of study drug.
* Male participants with a vasectomy must have had the vasectomy at least 90 days prior to randomization.
* Male participants must agree not to donate sperm from the Screening period through 90 days after the last dose.
* Understands the study procedures in the informed consent form and is willing and able to comply with the protocol
* Able to swallow tablets
* Supine blood pressure between 90/40 millimeters of mercury (mmHg) and 140/90 mmHg (inclusive) at Screening
* No clinically significant history or presence of ECG findings as judged by the PI at Screening and check-in, including each criterion as listed below:

  1. Normal sinus rhythm (heart rate between 45 beats per minute [bpm] and 100 bpm inclusive);
  2. Fridericia-corrected QTc (QTcF) interval < 450 milliseconds (msec);
  3. QRS interval ≤ 110 msec; and confirmed by manual over read if > 110 msec;
  4. PR interval ≤ 220 msec;
  5. No electrographically significant abnormalities that might interfere with ECG analysis including evidence of a previous myocardial infarction (MI), significant left ventricular hypertrophy (LVH), flat T-waves (particularly in the inferior leads) or more than minor non-specific ST-T wave changes
* Has serum potassium, calcium, and magnesium levels within the normal range at Screening

Exclusion Criteria:

* Participant is mentally or legally incapacitated or has significant emotional problems at the time of the Screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI
* History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the participant by their participation in the study
* History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose of study drug
* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs, related compounds, or inactive ingredients
* History of significant multiple and/or severe allergies (e.g., latex allergy, band aids, adhesive dressing, or medical tape), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs
* Female participants who are pregnant or lactating
* Positive urine drug or alcohol results at Screening or check-in
* Positive results at Screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Unable to refrain from or anticipates the use of:

  1. Any drug, including prescription and non-prescription medications (including antacids), herbal remedies, or vitamin supplements (especially those containing magnesium, aluminum, iron, or zinc) beginning 14 days prior to the first dose of study drug and throughout the study. Co-administration of ETX2514 and probenecid is prohibited.
  2. Any drugs known to be significant inhibitors or inducers of cytochrome P450 (CYP) enzymes and/or permeability glycoprotein (P-gp), including St. John's Wort, for 28 days prior to the first dose of study drug and throughout the study.
* Has been on a diet incompatible with the on-study diet (including an extreme diet which resulted in a significant weight change for whatever reason), in the opinion of the PI, within the 28 days prior to the first dose of study drug, and throughout the study
* Donation of blood or significant blood loss more than 500 milliliters (mL) within 56 days prior to the first dose of study drug
* Plasma donation within 7 days prior to the first dose of study drug
* Has had surgery or any medical condition which may affect the absorption, distribution, metabolism, or elimination of the study drug within 6 months prior to the first dose, in the opinion of the PI
* Participation in another clinical trial within 28 days prior to the first dose of study drug. The 28-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study.
* Participation in a previous clinical trial where participant received ETX2514
* History or presence of:

  1. hypokalemia, in the opinion of the PI;
  2. risk factors for Torsades de Pointes (e.g., heart failure, cardiomyopathy, or family history of Long QT Syndrome);
  3. sick sinus syndrome, second- or third-degree atrioventricular block, pulmonary congestion, cardiac arrhythmia, prolonged QT interval, or conduction abnormalities;
  4. repeated or frequent vasovagal episodes:

     * hypertension, angina, bradycardia, or severe peripheral arterial circulatory disorders;
     * history or evidence of any of the following: MI, cardiac valvulopathy, cardiac surgery revascularization (coronary artery bypass grafting or percutaneous transluminal coronary angioplasty), unstable angina, cerebrovascular accident or stroke or transient ischemic attack (TIA), pacemaker; atrial fibrillation, flutter, or non-sustained or sustained ventricular tachycardia (VT); pulmonary arterial hypertension; unexplained syncope or syncope within the last 3 years regardless of etiology; and/or history of hypokalemia
* Participant has a history within the last 6 months of frequent strenuous exercise, and/or is unwilling to refrain from strenuous exercise from 7 days prior to baseline Day -1 through the last Follow-Up Visit.
* Participants who refused to abstain from caffeine-containing foods or caffeinated beverages (e.g., coffee, tea, cola, energy drinks) for 7 days prior to Day -1 through the last Follow-up Visit
* Participants who refused to abstain from alcohol from 7 days prior to Day -1 through the last Follow-Up Visit
* Participants who refused to abstain from grapefruit-containing foods or beverages or Seville orange-containing foods or beverages from 2 weeks prior to Day -1 through the last Follow-Up Visit
* Participant has consumed cruciferous vegetables (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard greens) or charbroiled meats within 7 days prior to check-in through the last Follow-up Visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected change from Baseline in Fridericia-corrected QTc (QTcF) (ΔΔQTcF) | Baseline; up to Day 22

SECONDARY OUTCOMES:
Change from baseline in heart rate (HR) (ΔHR) | Baseline; up to Day 22
Change from Baseline in QTcF (ΔQTcF) | Baseline; up to Day 22
Change from Baseline in the PR interval (ΔPR) | Baseline; up to Day 22
Change from Baseline in the QRS interval (ΔQRS) | Baseline; up to Day 22
Placebo-corrected change from Baseline in HR (ΔΔHR) | Baseline; up to Day 22
Placebo-corrected change from Baseline in PR (ΔΔPR) | Baseline; up to Day 22
Placebo-corrected change from Baseline in QRS (ΔΔQRS) | Baseline; up to Day 22
Number of participants with categorical outliers for QTcF, HR, PR, and QRS | up to Day 22
Number of participants with treatment-emergent changes of T-wave morphology and U-wave presence | up to Day 22

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron Clinical Pharmacology Center, Baltimore, Maryland, United States